CLINICAL TRIAL: NCT03777592
Title: Correlation Between Perioperative Erector Spinae Plane Block and Postoperative Pain in Thoracoscopic Surgery
Brief Title: Perioperative Erector Spinae Plane Block in Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Sung Hyun Lee, Assistant Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-09-017-001
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Pain, Postoperative; Regional Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB with local agent (Active Comparator): ESPB will be performed using 20ml of 0.5% ropivacaine.
  Interventions: Procedure: erector spinae plane block
- ESPB with saline (Sham Comparator): ESPB will be performed using 20ml of saline.
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Procedure: erector spinae plane block — local anesthetic or saline is administered in to the interfascial plane between the transverse process of the vertebra and the erector spinae muscles, spreading to multiple paravertebral spaces

SUMMARY:
The erector spinae plane block (ESPB) is a novel myofascial plane block. The ESPB is targeted at anterior surface of the erector spinae plane, which is oriented cephalocaudally to the spinal transverse process. Local anaesthetic injected in this plane can block the dorsal rami and ventral rami and intercostal nerves. The aim of this study was to evaluate the effect of ESPB on postoperative pain in thoracic surgery.

DETAILED DESCRIPTION:
The erector spinae plane block (ESPB) is a newly defined regional anesthesia technique for thoracic analgesia. The blocks were performed at the T5 level of the spine using an in-plane approach.Previous studies were not designed as randomized controlled trial. In this study, the efficacy of ESPB is to confirm with randomized controlled trial design. ESPB will be performed in video assisted thoracoscopy preoperatively. After the surgery, the efficacy of ESPB will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Patients with physical class 1, 2
* Patients undergoing video assisted thoracoscopic surgery

Exclusion Criteria:

* Patients who experienced side effects on local anesthetics
* Patients with abnormal blood coagulation tests (INR> 1.5)
* Pregnant or lactating patients

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Pain scale | the first 5 min after arriving at the recovery room
  11-point numeric rating scale(
  (Scores from 0 to 10 are scored. The higher the score, the higher the degree of pain.The score is given in units of one point.)
Pain scale | 20 min after arriving at the recovery room
  11-point numeric rating scale (Scores from 0 to 10 are scored. The higher the score, the higher the degree of pain.The score is given in units of one point.)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Hyun Lee, MD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- KangbukSamsung Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No